CLINICAL TRIAL: NCT04568629
Title: Study of Advice and Decision-making on Prognosis Using the Judge-advisor System Within Multi-disciplinary Teams (ADJUST)
Brief Title: ADJUST: A Study on MDT Prognostication
Acronym: ADJUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17031/001
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-09

CONDITIONS: Terminal Illness
Keywords: Prognostication; Multidisciplinary teams; Judge-Advisor System; Palliative Care; End-of-life
MeSH Terms: conditions — Death

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two study arms and received advice reportedly from either a prognostic algorithm, or another clinician.
Who Masked: Participant, Investigator
Masking Description: The research team and participants were blind to intervention allocation, whilst the database specialist was not blinded to allocation. Group allocation was only revealed once the database had been locked and analyses had been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Algorithm Arm (Experimental): Participants received prognostic advice from a prognostic algorihm.
  Interventions: Other: Advice from the PiPS-B14 prognostic tool
- Clinician arm (Experimental): Participants recieved prognostic advice from another clinician.
  Interventions: Other: Advice from another clinician

INTERVENTIONS:
Other: Advice from the PiPS-B14 prognostic tool — Participants were informed that prognostic advice came from the PiPS-B14 prognostic tool. PiPS-B14 is a validated prognostic algorithm that has been shown to be as accurate as an agreed multi-professional survival estimate.
  Participants were further informed that in a previous study the PiPS-B14 risk categories for predicting two-week survival were as accurate as a doctor's or a nurse's prediction.
  Arms: Algorithm Arm
Other: Advice from another clinician — Participants were informed that prognostic advice came from another clinician.
  Doctors were told that advice was from a nurse, whereas nurses or other types of HCPs were told that advice was from a doctor.
  Arms: Clinician arm

SUMMARY:
This study investigates how clinicians form intuitive judgements about the prognoses of palliative care patients after receiving advice perceived as coming from either a team member or an algorithm.

DETAILED DESCRIPTION:
Using the Judge-Advisor System, the investigators will recruit clinicians working in palliative care for adults. Participants will be asked to complete an online survey and review five patient summaries ("vignettes") based on real cases derived from a previous study. Clinicians will be presented with key prognostic information and will be asked to provide an estimate of the probability that the patient will survive for two weeks (0-100%). After providing this initial estimate, participants will receive prognostic advice. While in reality all participants will receive the same advice, participants will be randomised into two groups and these groups will be informed that the advice is either: (1) provided by an algorithm; or (2) provided by a team colleague. Participants will then be given the opportunity to give a second, possibly revised estimate in the light of the advice received.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians working in an adult palliative care service
* Willing and able to provide written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Probability of survival estimate | Participants will have up to 7 months (until the study closes) to provide an estimate for each vignette
  Clinicians' estimates of the probability of a patient surviving for two weeks (0-100%)

SECONDARY OUTCOMES:
Participants' weighting policies (characteristics of the participants) | Participants will have up to 7 months (until the study closes) to provide an estimate for each vignette
  Participants' responses to demographic questions
Participants' weighting policies (the advice itself) | Participants will have up to 7 months (until the study closes) to provide an estimate for each vignette
  Strength of the prognostic advice provided by the advisor (0-100%)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stone, MA MD FRCP, Principal Investigator — UCL (University College London)
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data (suitably anonymised) may be shared with other research groups if a reasonable request is submitted to and agreed by the CI
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after the publication of results and will be archived securely by the Chief Investigator for a minimum of 20 years from the declaration of end of study
Access Criteria: The data will be shared upon reasonable request

REFERENCES:
- [Derived] Bruun A, White N, Oostendorp L, Vickerstaff V, Harris AJL, Tomlinson C, Bloch S, Stone P. An online randomised controlled trial of prognosticating imminent death in advanced cancer patients: Clinicians give greater weight to advice from a prognostic algorithm than from another clinician with a different profession. Cancer Med. 2023 Mar;12(6):7519-7528. doi: 10.1002/cam4.5485. Epub 2022 Nov 29. PMID 36444695

DOCUMENTS (2):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT04568629/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT04568629/SAP_000.pdf